CLINICAL TRIAL: NCT02737124
Title: Prospective Randomized Control Trial Assessing Effects of Pre-Operative Acetaminophen in Isolated Meniscectomy Patients
Brief Title: Acetaminophen Randomized Controlled Trial
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is currently Lapsed
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01297
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Post Operative Pain
Keywords: Acetaminophen; Surgery; Meniscectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1000 Mg Acetaminophen (Experimental): Acetaminophen will be given 24 hours before surgery
  Interventions: Drug: Acetaminophen
- Placebo (Active Comparator): A sugar pill will be given 24 hours before the scheduled surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen will be given 24 hours before scheduled surgery.
  Arms: 1000 Mg Acetaminophen
Other: Placebo — Placebo will be given to subjects 24 hours before scheduled surgery.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Patients that are to undergo isolated meniscectomy will be randomized to 2 cohorts: one will take the FDA recommended dose of acetominophen (1000mg) 24hrs before surgery, one will be given a similarly looking placebo pill. A multitude of post-op variables will be included, mainly pain scores and morphine equivalent doses at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* ASA Class I-II
* Patients scheduled for meniscectomy

Exclusion Criteria:

* Contraindication to acetaminophen (hypersensitivity, extensive alcohol history, liver disease, actively breastfeeding)
* Legally incompetent or mentally impaired (e.g., minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age or older than 65
* Any patient considered a vulnerable subject
* Patients on pain medication prior to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Morphine-equivalent dose consumption | 7 days
  Total morphine-equivalent dose consumption during immediate post-op, phase 1 recover, phase II recovery, at 2 days, and at 7 days
Pain using the visual analogue scale | 7 Days
  The visual analogue scale is a scale with a line from 0 on one side and 100 on the other where the patient is asked to mark where they believe their pain is.
Narcotic Use | 7 Days
  Total morphine-equivalent dose consumption during immediate post-op, phase 1 recover, phase II recovery, at 2 days, and at 7 days will also be recorded.
Measure of time to discharge from the PACU | 7 Days
  Time to discharge from the PACU
Measure of time to discharge from hospital | 7 Days
  Time to discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States